CLINICAL TRIAL: NCT01448447
Title: Phase IV Trial to Evaluate Breast Brachytherapy Using the Mammosite-Ml® Radiation Therapy Delivery System as the Sole Method of Radiation Therapy or as a Boost for Early Stage Breast Cancer and Ductal Carcinoma In Situ of the Breast
Brief Title: Phase IV Trial to Evaluate Breast Brachytherapy Using the Mammosite-Ml®
Acronym: Mammosite ML
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Research (Other)
Responsible Party: Principal Investigator, Robert Frazier, MD, MD, Radiation Oncologist, Mercy Research
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mammosite ML
Record Dates: First submitted 2011-09-30; First posted 2011-10-07 (Estimated); Results first posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer; Ductal Carcinoma in Situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sole method (Experimental): patients will be treated with HDR brachytherapy using Mammosite ML as the sole method for radiation delivery after lumpectomy for breast cancer or DCIS
  Interventions: Device: Mammosite ML
- Boost (Experimental): patients will be treated with HDR brachytherapy using Mammosite ML as a boost technique prior to standard external beam radiation after lumpectomy for breast cancer or DCIS
  Interventions: Device: Mammosite ML

INTERVENTIONS:
Device: Mammosite ML — 34 Gy / 10 fractions (3.4 Gy per fraction) 2 fractions / day (separated by at least 6 hours) Delivered in 5 consecutive working days
  Other Names: HDR Brachytherapy
  Arms: Sole method
Device: Mammosite ML — 5-10.2 Gy / 2-3 fractions (3.4 Gy per fraction) 2 fractions / day (separated by at least 6 hours) Delivered in 1-2 days Followed by whole breast radiation (25-28 daily tx)
  Other Names: HDR Brachytherapy
  Arms: Boost

SUMMARY:
This study will evaluate the local control rate, cosmetic results, and complication rates of breast brachytherapy delivered using the MammoSite-ML® when used as the sole method of radiation therapy or as a boost technique for patients with stage I-II carcinoma of the breast (< 3 cm), (non-lobular histology) treated with lumpectomy with histologically negative surgical margins by at least 2 mm, negative axillary lymph nodes, and DCIS.

Hypotheses:

* For selected patients with stage I breast carcinoma and Ductal Carcinoma In Situ (DCIS), radiation therapy delivered with brachytherapy alone using the MammoSite-ML® is technically feasible and reproducible with acceptable complication rates.
* Cosmetic results after brachytherapy will be similar to that obtained after traditional whole breast external beam radiation therapy.
* Local tumor control rate in the breast after brachytherapy will be similar to that of conventional external beam radiation therapy, with less inconvenience and potentially less cost to the patient, given the selection criteria which minimize the risk of clinically significant multicentric or extensive residual carcinoma following lumpectomy.

ELIGIBILITY:
Inclusion Criteria:

* Women,age of at least 45 years
* Zubrod performance status of 0-2
* AJCC Stage I-II (T1-T2, N0 M0) breast cancer
* Maximum tumor dimension < 3 cm
* Invasive ductal, medullary, papillary, tubular, colloid (mucinous) histologies
* Unifocal breast cancer
* Unilateral breast cancer (no synchronous or previous contralateral breast cancer)
* Lumpectomy with negative surgical margins by at least 2 mm or re-excision specimen with negative surgical margins by at least 2 mm
* Ductal Carcinoma In-Situ
* Negative axillary lymph nodes for invasive breast cancer (sentinel node biopsy or standard level I-II dissection with > 6 nodes removed)
* Time interval from final breast surgery to brachytherapy loading less than 8 weeks
* At least 2 mm of breast tissue between the skin and the MammoSite® balloon surface(prefer > 5 mm)
* If chemotherapy is planned, it must begin no earlier that 2 weeks following completion of radiation therapy. If chemotherapy is first, a minimum of 2 weeks from the last cycle must elapse prior to the start of radiation therapy.
* Signed study-specific consent form

Exclusion Criteria:

* Invasive lobular histology
* Non-epithelial breast malignancies such as sarcoma or lymphoma
* Multifocal or multicentric invasive carcinoma
* Extensive intraductal component (EIC)
* Paget's disease of the nipple
* Skin involvement by tumor, regardless of tumor size
* Positive axillary lymph nodes
* Distant metastases
* Collagen vascular disease (scleroderma)
* Pregnant or lactating women, due to potential exposure of the fetus to RT and unknown effects of RT on lactating females (negative pregnancy test for women of child-bearing age)
* Any previously treated or synchronous contralateral breast carcinoma
* Patients with psychiatric or addictive disorder that would preclude obtaining informed Consent
* Men

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-12; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bethany G Sleckman, MD, Principal Investigator — Mercy Hospital St. Louis
Locations (2):
- United States (2):
  - Mercy Clinic St. Louis Cancer and Breast Institute, St Louis, Missouri
  - Mercy Hospital St. Louis, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sole Method | Boost
Started | 20 | 0
Completed | 20 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 20 patients were enrolled within sole method arm, no patients were enrolled in boost method arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Sole Method | Boost | Total
Number analyzed (Participants) | 20 | 0 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 6 |  | 6
  >=65 years | 14 |  | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 |  | 20
  Male | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Ipsilateral Recurrence Rate
Description: * Local recurrence is defined as either invasive or non-invasive breast cancer recurrence within the target volume.
  * Elsewhere recurrence is defined as either invasive or non-invasive breast cancer recurrence outside of the target volume.
  * Local control rate will be evaluated by imaging techniques, physical exam and biopsy, if applicable.
  Measured as a count of participants experiencing recurrence, i.e. each subject experiencing ipsilateral tumor recurrence within 5 years = 1, and each subject with no ipsilateral tumor recurrence within 5 years = 0
Time Frame: 5 years
Population: 11 patients within sole method arm were lost to follow-up prior to 5 year follow-up period.
Measure: Number; unit: participants
Arm/Group | Sole Method | Boost
Number analyzed (Participants) | 9 | 0
participants | 0 |

2. Secondary Outcome: Cosmetic Results
Description: Evaluation of cosmetic results as judged by the patient, surgeon, and radiation oncologist at stated follow up intervals. Serial photographs will be obtained. The cosmetic results will be assessed using the four category Harvard Scale definitions: Excellent - The treated breast looks essentially the same as the opposite breast Good - Minimal but identifiable effects of radiation on the treated breast Fair - Significant effects of radiation on the treated breast Poor - Severe normal tissue sequelae secondary to irradiation
Time Frame: 6 months after treatment, then annually for 5 years
Population: No patient information was collected for boost method arm as no patients were enrolled into boost method arm.
  11 participants in sole method arm were lost to follow-up over 5 year period.
Measure: Count of Participants; unit: Participants
Arm/Group | Sole Method | Boost
Number analyzed (Participants) | 20 | 0
Participants
  Number of pts with "excellent" cosmetic results, 1 year post treatment | 4 | 0
  Number of pts with "good" cosmetic results, 1 year post treatment | 14 | 0
  Number of pts with "fair" cosmetic results, 1 year post treatment | 0 | 0
  Number of pts with "poor" cosmetic results, 1 year post treatment | 0 | 0
  Number of pts with "excellent" cosmetic results, 2 years post treatment | 4 | 0
  Number of pts with "good" cosmetic results, 2 years post treatment | 12 | 0
  Number of pts with "fair" cosmetic results, 2 years post treatment | 0 | 0
  Number of pts with "poor" cosmetic results, 2 years post treatment | 0 | 0
  Number of pts with "excellent" cosmetic results, 3 years post treatment | 4 | 0
  Number of pts with "good" cosmetic results, 3 years post treatment | 10 | 0
  Number of pts with "fair" cosmetic results, 3 years post treatment | 0 | 0
  Number of pts with "poor" cosmetic results, 3 years post treatment | 0 | 0
  Number of pts with "excellent" cosmetic results, 4 years post treatment | 4 | 0
  Number of pts with "good" cosmetic results, 4 years post treatment | 8 | 0
  Number of pts with "fair" cosmetic results, 4 years post treatment | 0 | 0
  Number of pts with "poor" cosmetic results, 4 years post treatment | 0 | 0
  Number of pts with "excellent" cosmetic results, 5 years post treatment | 3 | 0
  Number of pts with "good" cosmetic results, 5 years post treatment | 6 | 0
  Number of pts with "fair" cosmetic results, 5 years post treatment | 0 | 0
  Number of pts with "poor" cosmetic results, 5 years post treatment | 0 | 0

3. Secondary Outcome: Toxicity Measured Through Adverse Event Incidence
Description: The incidence of serious adverse events will be calculated. Adverse events reviewed for device harm/toxicity include skin redness, breast pain, infections, breast swelling, and rib fractures.
Time Frame: during therapy, 6 weeks after completion of therapy, and additionally as needed
Population: No patient information was collected for boost method arm as no patients were enrolled into boost method arm of study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sole Method | Boost
Number analyzed (Participants) | 20 | 0
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events will be collected during follow-up visits non-systematically over the course of 5 years beginning from procedure.
Description: Adverse event information not collected from boost method arm patients, as there were no patients enrolled for the boost method arm.
Arm/Group | Sole Method | Boost
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/0
Other Adverse Events (participants affected / at risk) | 1/20 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sole Method (N=20) | Boost (N=0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No